CLINICAL TRIAL: NCT03110445
Title: Monocentric Open Label Phase I Immunotherapy Trial of Breast Cancer Patients With a Non-replicating Recombinant Vaccinia Virus Expressing Cancer/Testis Antigens and Cluster of Differentiation Antigen 80 (CD80)-CD40L Costimulatory Molecules.
Brief Title: Cancer/Testis Antigen Immunotherapy Phase I Study With 740-CTA Vaccinia Virus
Acronym: rVV-740CTA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: not sufficiently staff available to perform trial
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKNZ 2015-026
Record Dates: First submitted 2016-05-11; First posted 2017-04-12 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rVV-740CTA vaccine (Experimental)
  Interventions: Biological: rVV-740CTA

INTERVENTIONS:
Biological: rVV-740CTA — non replicating recombinant vaccinia virus expressing 7 Cancer Testis Antigen (CTA) epitopes together with CD80 and CD154(40L)

SUMMARY:
Monocentric open-label phase I/II trial aiming at evaluating, in adjuvant setting, safety (primary outcome), immunological and clinical efficacy (secondary outcomes) of a non replicating recombinant vaccinia virus expressing cancer/testis antigen (CTA) derived epitopes and CD80 and CD40 ligand (CD40L, CD154) costimulatory molecules in patients with CTA expressing tumors.

ELIGIBILITY:
Inclusion Criteria:

* Surgically treated M0 patients with solid tumors
* Tumor expressing at least one of the vaccine targeted antigens Melanoma-associated antigen (MAGE)-A1, -A2,
* A3, -A4, -A6, -A10, -A12 or New York (NY) esophageal squamous cell carcinoma-1 (ESO-1) (NY-ESO-1) (by real-time quantitative PCR (RT-qPCR))
* Patient expressing the targeted Human Leukocyte Antigen (HLA) restriction (A0201 /A0101/ B3501)
* 4 weeks interval following surgical resection of tumor and, if applicable, completion of adjuvant therapy.
* Karnofsky over 70%
* No other concomitant malignancy

Exclusion Criteria:

* History of anaphylaxis or severe allergic reaction
* Severe heart, lung, kidney, liver or psychiatric condition
* Concurrent immunosuppressive therapy or impaired immune system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
number of adverse Events | 2 years
  Safety measured by assessment of number of adverse events that have occured
number of serious adverse Events | 2 years
  Safety measured by assessment of number of serious adverse Events that have occured

SECONDARY OUTCOMES:
Evolution of Immune reactivity to the CTA | 18 months
  Vaccine epitopes specific CD8+ T-cell responses will be evaluated from peripheral blood samples prior, during and after treatment.
Disease free survival | 2 years
  number of patients with no relapse of disease at timepoint 2 years
Overall survival | 2 years
  number of patients still living at timepoint 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul ZAJAC, PhD, Study Director — University Hospital Basel - Dept of Biomedicine; Walter WEBER, MD, Principal Investigator — University Hospital of Basel - Dept of Surgery

IPD SHARING:
Plan to Share IPD: No
publication per reviewed journal